CLINICAL TRIAL: NCT05202860
Title: Impact of Human Papillomavirus (HPV) Vaccination on Burden of Disease in Patients with Actinic Keratosis - a Double-blind Randomized Controlled Trial
Brief Title: Impact of Human Papillomavirus (HPV) Vaccination on Burden of Disease in Patients with Actinic Keratosis
Acronym: VAXAK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Sponsor-Investigator, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2021-003895-15; H-21047863 (Other: National Committee on Health Research Ethics (NVK; Denmark))
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Actinic Keratoses; Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Basal Cell; Carcinoma, Squamous Cell | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPV vaccine (Experimental): Commercially available nonavalent HPV vaccine (Gardasil(R) 9) given intramuscularly at baseline, month 2 and month 6
  Interventions: Biological: HPV Vaccine
- Isotonic Saltwater Vaccine (Placebo Comparator): 0.9% NaCl given intramuscularly at baseline, month 2 and month 6
  Interventions: Biological: PLACEBO vaccine

INTERVENTIONS:
Biological: HPV Vaccine — (Gardasil 9 human papilloma vaccine)
  Arms: HPV vaccine
Biological: PLACEBO vaccine — Isotonic saltwater sham vaccine
  Arms: Isotonic Saltwater Vaccine

SUMMARY:
A double-blind, randomized, placebo controlled intervention trial on patients with actinic keratosis.

DETAILED DESCRIPTION:
Endeavoring to develop a new therapeutic and preventative strategy for patients with AK, this study aims to investigate the impact of 9-valent HPV vaccination on AK burden and -development over the course of 12 months.

Seventy actinic keratosis (AK) patients are randomized 1:1 to two parallel groups that receive blinded HPV vaccination or sham placebo (isotonic NaCl) vaccination at baseline (day 0), month 2 and month 6. At month 6 and 9, both groups undergo lesion-directed cryotherapy of Olsen grade II-III AKs. Treatment response, based on percentage change (%) in baseline number of AK lesions in a predefined test area (primary outcome), is evaluated at months 2, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria are eligible to participate in this study:

1. High AK burden, defined as ≥15 AK lesions in the included test area (50-100 cm2) at baseline
2. Test area does not involve the ala nasi, eyelids, nasolabial folds, or periauricular skin
3. >18 years of age at baseline
4. Fitzpatrick skin phototype I-IV
5. Legally competent, able to give verbal and written informed consent
6. Subject is willing to participate and can comply with protocol requirements including the refraining from other therapy (with the exception of KC treatment) in the test area for the duration of the trial.
7. Women of childbearing potential1 must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment and be on effective contraception2 until discontinuation of the vaccine therapy. Additional pregnancy testing will not be conducted unless pregnancy is suspected.

1Female subjects are considered of childbearing potential unless they have been hysterectomized or have undergone tubal ligation or have been post-menopausal for at least one year prior to first visit.

2Intrauterine device or hormonal contraception (oral, implant, patch, vaginal ring, injection).

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible to participate in this study:

1. Known or suspected immunosuppression (by disease or immunosuppressive drug)
2. History of vaccine-related allergic reactions or known allergy to Gardasil®9 ingredients or yeast
3. Previously vaccinated with any HPV vaccine
4. History of keloids
5. Other skin diseases present in the test area at baseline
6. Lactating or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2034-06-19 (Estimated)

PRIMARY OUTCOMES:
Treatment response in HPV vaccinated versus control group | Evaluated at month 2, 6, 9, and 12
  Percentage change from baseline (%) in number of AK lesions (grades I and II-III) in the selected test area

SECONDARY OUTCOMES:
New AK lesions | Evaluated at month 2, 6, 9, 12
  New AK lesions (n) arising in the test area since last visit
Partial (≥75%) clearance | Evaluated at month 12
  Atleast 75 % reduction in total number of AK lesions compared to baseline
Complete (100%) clearance | Evaluated at month 12
  100% reduction in total number of AK lesions compared to baseline
Side Effects | Evaluated over the course of 12 months
  Occurence of local and systemic side effects in HPV vaccinated versus control group
New Keratinocyte Carcinomas (KCs) | Evaluated at month 2, 6, 9, and 12
  New KCs (basal or squamous cell carcinoma) identified anywhere on the body of participants in HPV vaccinated versus control group registered over the course of the 12-month trial, compared to average yearly whole-body KC rate (determined by assessment of electronic medical record/patobank results) up to 3 years prior to baseline.
Long term Keratinocyte Carcinoma (KC) rates | 10 years
  Annual rate and total number of histologically confirmed KC lesions determined by assessment of electronic medical record/patobank results assessed 3, 5 and 10 years after vaccination compared to KC rates up to 5 years prior to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, PhD, DMSc, Principal Investigator — Bispebjerg Hospital; Emily Wenande, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wenande E, Hastrup A, Wiegell S, Philipsen PA, Thomsen NB, Demehri S, Kjaer SK, Haedersdal M. Human Papillomavirus Vaccination and Actinic Keratosis Burden: The VAXAK Randomized Clinical Trial. JAMA Dermatol. 2025 Jun 1;161(6):605-614. doi: 10.1001/jamadermatol.2025.0531. PMID 40047786